CLINICAL TRIAL: NCT05132855
Title: Safety, Reactogenicity, and Immunogenicity of Heterologous Boost Third Dose of mRNA and Protein COVID-19 Vaccine: a Single-blind and Randomized Study
Brief Title: The Immune Response of Heterologous Boost Third Dose of mRNA and Protein COVID-19 Vaccine
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Medigen Vaccine Biologics Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 202101767A3
Record Dates: First submitted 2021-11-11; First posted 2021-11-24 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2021-11

CONDITIONS: COVID-19; Breakthrough Infection
Keywords: COVID-19; Breakthrough infection; Heterologous vaccine booster; mRNA vaccine; Protein subunit vaccine
MeSH Terms: conditions — COVID-19; Breakthrough Infections | interventions — BNT162 Vaccine; 2019-nCoV Vaccine mRNA-1273; MVC-COV1901 vaccine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Booster group 1 (BNT162b2 30ug) (Experimental): The participants in this group will receive BNT162b2 30ug as the booster dose.
  Interventions: Biological: BNT162b2
- Booster group 2 (mRNA-1273 50ug) (Experimental): The participants in this group will receive mRNA-1273 50ug as the booster dose.
  Interventions: Biological: mRNA-1273
- Booster group 3 (mRNA-1273 100ug) (Experimental): The participants in this group will receive mRNA-1273 100ug as the booster dose.
  Interventions: Biological: mRNA-1273
- Booster group 4 (MVC-COV1901 15ug) (Experimental): The participants in this group will receive MCV COVID-19 vaccine 15ug as the booster dose.
  Interventions: Biological: MVC-COV1901

INTERVENTIONS:
Biological: BNT162b2 — BNT162b2 is an mRNA vaccine to prevent COVID-19 infection and is approved by the emergency use of authorization (EUA) by the Taiwan FDA.
  Arms: Booster group 1 (BNT162b2 30ug)
Biological: mRNA-1273 — mRNA-1273 is an mRNA vaccine to prevent COVID-19 infection and is approved by the emergency use of authorization (EUA) by the Taiwan FDA.
  Arms: Booster group 2 (mRNA-1273 50ug); Booster group 3 (mRNA-1273 100ug)
Biological: MVC-COV1901 — MCV COVID-19 vaccine is a protein subunit vaccine containing S2P S-protein which passes the EUA by Taiwan FDA.
  Arms: Booster group 4 (MVC-COV1901 15ug)

SUMMARY:
The severe acute respiratory syndrome coronavirus 2 (SARS-COV-2) specific antibody and neutralizing antibody level induced by adenovirus vector vaccines were lower than mRNA vaccines. Vaccine efficacy of ChAdOx1 nCoV-19 was lower than BNT162b2 and mRNA 1273 in clinical trials. The emergence of highly transmissible and mutant variants of SARS-COV-2 has raised the concern of COVID-19 vaccine effectiveness. The complete vaccination rate is still low in Taiwan. Strict border control measures are imposed by Central Epidemic Command Center. However, the measure of quarantine for flight crew is considered one of the breach of COVID-19 infection control. Despite most of the flight crew has fully vaccinated, several episodes of breakthrough infection occurred among flight crew resulting in domestic infection recently. Low neutralizing antibody was found in a proportion of fully vaccinated flight crew and healthcare workers. A 3rd booster COVID-19 dose is considered for flight crew and healthcare workers. This study is to determine the safety, reactogenicity, and immunogenicity of heterologous 3rd booster of mRNA and protein COVID-19 vaccines.

DETAILED DESCRIPTION:
Safety concerns of COVID-19 ChAdOx1 nCoV-19 vaccine have led to a recommendation of heterologous boost with mRNA vaccine in several countries. Initial safety data of heterologous prime-boost with ChAdOx1 nCoV-19 and BNT162b2 vaccines showed well-tolerated. No major differences in reactogenicity were observed between homologous and heterologous vaccination. Immunogenicity of heterologous ChAdOx1 nCoV-19 and BNT162b2 vaccination is better compared with homologous ChAdOx1 nCoV-19 vaccination. Despite the scarcity of safety and immunogenicity of heterologous ChAdOx1 nCoV-19 and mRNA 1273 vaccination, the preliminary reports revealed similar findings. Although both T and B memory cells contribute to the protection, there is evidence that neutralizing serum antibody levels have high correlates of protection for symptomatic SARS-COV-2 infection. The SARS-COV-2 specific antibody and neutralizing antibody level induced by adenovirus vector vaccines were lower than mRNA vaccines. Vaccine efficacy of ChAdOx1 nCoV-19 was lower than BNT162b2 and mRNA 1273 in clinical trials. In the real world, the ChAdOx1 nCoV-19 vaccine appeared less effective than the BNT162b2 and mRNA1273 vaccine in preventing SARS-COV-2 infection. The emergence of highly transmissible and mutant variants of SARS-COV-2 has raised the concern of COVID-19 vaccine effectiveness. The S protein of the widespread SARS-COV-2 delta variant reduced the binding of neutralizing antibodies. Breakthrough infections are increasing worldwide. Vaccine effectiveness decreased significantly after the emergence of the SARS-COV-2 delta variant. Waning immunity is another potential cause of breakthrough infection. Centers for Disease Control of the United States has advocated 3rd booster dose of mRNA vaccine for people at risk of COVID-19 and those who work in high-risk settings including healthcare workers. Israel expanded its 3rd COVID-19 vaccine boost to those aged over 12 years old. The complete vaccination rate is still low in Taiwan. Strict border control measures are imposed by Central Epidemic Command Center. However, the measure of quarantine for flight crew is considered one of the breaches of COVID-19 infection control. Despite most of the flight crew has fully vaccinated, several episodes of breakthrough infection occurred among flight crew resulting in domestic infection recently. Low neutralizing antibody was found in a proportion of fully vaccinated flight crew and healthcare workers. A 3rd booster COVID-19 dose is considered for flight crew and healthcare workers. This study is to determine the safety, reactogenicity, and immunogenicity of heterologous 3rd booster of mRNA and protein COVID-19 vaccines.

With waning vaccine induced immunity and emergence of potent immune evasion SARS-CoV-2 omicron variant, previous virus and vaccine-induced immunity have failed to prevent transmission. Build-up of herd immunity through vaccination is no longer achievable so far. On the other hand, SARS- CoV-2 omicron induced immunity has been shown low cross-protective against other variants. Omicron breakthrough infection can boost existing immunity induced by vaccination. The neutralizing titer elicited by omicron breakthrough infection are much higher than that induced by 3 doses of mRNA vaccines. Hybrid immunity by vaccination and omicron breakthrough infection can elicit effective cross-neutralizing antibodies against most variants.

More than 10% of population in Taiwan have infected with omicron variant. Second booster vaccination is being advocated for health care workers. The study of dynamics of immunogenicity induced by third dose heterologous booster vaccination needs to be revised. Immunogenicity including SARS-CoV-2 anti- spike IgG, the 50% neutralizing antibody titer and IFN-secreting T cells specific to whole spike protein will be performed at 180 days after booster vaccination as schedule. Additional memory T cell epitopes and memory B cell epitopes will be studied. Some participants have been infected with the omicron variant. We will compare differences of memory T cell epitopes and memory B cell epitopes between uninfected participants and omicron breakthrough infected participants. Besides, second booster vaccination is planning to be administered in health care workers. We will compare differences of memory T cell epitopes and memory B cell epitopes between 2 boosters vaccinated participants and SARS-CoV-2 breakthrough infected participants. Immunogenicity study will be conducted 28 days after the second booster vaccination and 28 days after SARS-CoV-2 breakthrough infection. Immunogenicity study, including SARS-CoV-2 anti- spike IgG, the 50% neutralizing antibody titer (NT50) and IFN-secreting T cells specific to whole spike protein, will be compared between participants with 2 booster vaccination and SARS-CoV-2 breakthrough infection.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is willing to give written informed consent for participation in the trial.
2. Participants should receive 2 doses of the AZD1222. Evidence of this will be gathered from medical history and/or medical records including the COVID-19 vaccine registration yellow card.

Exclusion Criteria:

The participant may not enter the trial if ANY of the following apply:

1. Fever or evidence of upper respiratory tract infections
2. Confirmed COVID-19 cases (PCR-confirmed infection or detectable anti-nucleocapsid protein IgG)
3. History of anaphylaxis, severe allergic disease, or reactions likely to be exacerbated by any component of study vaccines (e.g. hypersensitivity to the active substance or any of the listed ingredients of any study vaccine).
4. Malignancy requiring receipt of immunosuppressive chemotherapy or radiotherapy for treatment of solid organ cancer/hematological malignancy within the 6 months prior to enrollment.
5. Bleeding disorder (e.g. factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following intramuscular injections or venipuncture.
6. Has received vaccines other than COVID-19 vaccine within one month
7. Pregnancy or willingness/intention to become pregnant within 3 months post booster vaccine
8. Aged < 20 years or unable to sign the informed consent
9. Any other significant disease, disorder, or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study, or impair interpretation of the study data or insufficient level of language to undertake all study requirements in the opinion of the Investigators.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
The immune response after heterologous boost third dose of COVID-19 vaccines after homologous prime-boost AZD1222 vaccination | Day 28 after third dose boost
  Immunogenicity studies include SARS-CoV-2 anti-spike IgG, the 50% neutralizing antibody titer (NT50) and IFN - secreting T cells specific to whole spike protein.
The immune response after heterologous boost third dose of COVID-19 vaccines after homologous prime-boost AZD1222 vaccination | Day 180 after third dose boost
  Immunogenicity studies include SARS-CoV-2 anti-spike IgG, the 50% neutralizing antibody titer (NT50), IFN - secreting T cells specific to whole spike protein, and Memory T cell epitopes and memory B cell epitopes by flow cytometry.
The immune response after heterologous boost fourth dose of COVID-19 vaccines after homologous prime-boost AZD1222 vaccination | Day 28 after second booster vaccination.
  Immunogenicity studies include SARS-CoV-2 anti-spike IgG, the 50% neutralizing antibody titer (NT50), IFN - secreting T cells specific to whole spike protein, and Memory T cell epitopes and memory B cell epitopes by flow cytometry.
The immune response of breakthrough infection after heterologous boost third dose of COVID-19 vaccines after homologous prime-boost AZD1222 vaccination | Day 28 after breakthrough infection (after receiving third doses of any COVID-19 vaccine)
  Immunogenicity studies include SARS-CoV-2 anti-spike IgG, the 50% neutralizing antibody titer (NT50), IFN - secreting T cells specific to whole spike protein, and Memory T cell epitopes and memory B cell epitopes by flow cytometry.

SECONDARY OUTCOMES:
The safety of heterologous boost third dose of COVID-19 vaccines | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Evaluation of the safety profile included Solicited local adverse events (AEs), solicited systemic AEs, AE of special interest (AESI), and serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Hsun Chiu, MD, PhD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hillus D, Schwarz T, Tober-Lau P, Vanshylla K, Hastor H, Thibeault C, Jentzsch S, Helbig ET, Lippert LJ, Tscheak P, Schmidt ML, Riege J, Solarek A, von Kalle C, Dang-Heine C, Gruell H, Kopankiewicz P, Suttorp N, Drosten C, Bias H, Seybold J; EICOV/COVIM Study Group; Klein F, Kurth F, Corman VM, Sander LE. Safety, reactogenicity, and immunogenicity of homologous and heterologous prime-boost immunisation with ChAdOx1 nCoV-19 and BNT162b2: a prospective cohort study. Lancet Respir Med. 2021 Nov;9(11):1255-1265. doi: 10.1016/S2213-2600(21)00357-X. Epub 2021 Aug 13. PMID 34391547
- [Background] Liu X, Shaw RH, Stuart ASV, Greenland M, Aley PK, Andrews NJ, Cameron JC, Charlton S, Clutterbuck EA, Collins AM, Dinesh T, England A, Faust SN, Ferreira DM, Finn A, Green CA, Hallis B, Heath PT, Hill H, Lambe T, Lazarus R, Libri V, Long F, Mujadidi YF, Plested EL, Provstgaard-Morys S, Ramasamy MN, Ramsay M, Read RC, Robinson H, Singh N, Turner DPJ, Turner PJ, Walker LL, White R, Nguyen-Van-Tam JS, Snape MD; Com-COV Study Group. Safety and immunogenicity of heterologous versus homologous prime-boost schedules with an adenoviral vectored and mRNA COVID-19 vaccine (Com-COV): a single-blind, randomised, non-inferiority trial. Lancet. 2021 Sep 4;398(10303):856-869. doi: 10.1016/S0140-6736(21)01694-9. Epub 2021 Aug 6. PMID 34370971
- [Background] Normark J, Vikstrom L, Gwon YD, Persson IL, Edin A, Bjorsell T, Dernstedt A, Christ W, Tevell S, Evander M, Klingstrom J, Ahlm C, Forsell M. Heterologous ChAdOx1 nCoV-19 and mRNA-1273 Vaccination. N Engl J Med. 2021 Sep 9;385(11):1049-1051. doi: 10.1056/NEJMc2110716. Epub 2021 Jul 14. No abstract available. PMID 34260850
- [Derived] Chuang CH, Huang CG, Huang CT, Chen YC, Kung YA, Chen CJ, Chuang TC, Liu CC, Huang PW, Yang SL, Gu PW, Shih SR, Chiu CH. Titers and breadth of neutralizing antibodies against SARS-CoV-2 variants after heterologous booster vaccination in health care workers primed with two doses of ChAdOx1 nCov-19: A single-blinded, randomized clinical trial. J Clin Virol. 2022 Dec;157:105328. doi: 10.1016/j.jcv.2022.105328. Epub 2022 Nov 12. PMID 36399969